CLINICAL TRIAL: NCT04298814
Title: Analysis of Safety Related Factors of Endotracheal Intubation in Patients With Severe Covid-19 Pneumonia
Brief Title: Safety Related Factors of Endotracheal Intubation in Patients With Severe Covid-19 Pneumonia
Status: Withdrawn | Type: Observational
Why Stopped: It was repeated with other studies in the same department
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, aijun xu, associate professor, Tongji Hospital
Other Study IDs: COVEI
Record Dates: First submitted 2020-02-26; First posted 2020-03-06 (Actual); Last update posted 2020-07-20 (Actual); Status verified 2020-07

CONDITIONS: COVID-19; Endotracheal Intubation
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: severe covid-19 pneumonia with ET — severe covid-19 pneumonia undergoing endotracheal intubation

SUMMARY:
To analyze the intubation with severe covid-19 pneumonia, the infection rate of anesthesiologist after intubation, and summarizes the experience of how to avoid the infection of anesthesiologist and ensure the safety of patients with severe covid-19 pneumonia.

DETAILED DESCRIPTION:
To analyze the intubation time, intubation condition, intubation process, intubation times and success rate of patients with severe covid-19 pneumonia, the infection rate of anesthesiologist after intubation, the degree of respiratory improvement and survival rate of patients, and summarizes the experience of how to avoid the infection of anesthesiologist and ensure the safety of patients with severe covid-19 pneumonia.

ELIGIBILITY:
Inclusion Criteria:

* Wuhan residents;
* novel coronavirus pneumonia was found to be characterized by fever and cough. Laboratory tests revealed leukocyte or lymphocyte decrease, chest CT examination showed viral pneumonia changes, and was diagnosed as COVID-19 pneumonia according to the national health and Health Committee's new coronavirus pneumonia diagnosis and treatment plan (trial version fifth Revision).
* Severe and critical patients with covid-19 pneumonia in urgent need of tracheal intubation;
* Sign informed consent.

Exclusion Criteria:

* Suspected patients with covid-19 pneumonia;
* Patients who need emergency endotracheal intubation due to other causes of respiratory failure;
* The family refused to sign the informed consent.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Severe and critical patients with covid-19 pneumonia in urgent need of tracheal intubation
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-08-07 (Estimated); Primary Completion 2020-12-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Success rate of intubation | the time span between 1hour before intubation and 24h after intubation
  The data of Success rate of intubation with severe COVID-19 pneumonia patients
Infection rate of Anesthesiologist | the time span between 1hour before intubation and 14days after intubation
  Infection rate of Anesthesiologist who performed the endotracheal intubation for severe COVID-19 pneumonia patients

SECONDARY OUTCOMES:
Extubation time | the time span between 1hour before intubation and 30days after intubation
  Extubation time of intubated severe COVID-19 pneumonia patients

CONTACTS AND LOCATIONS:
Overall Officials: Aijun XU, Dr., Principal Investigator — Tongji Hospital
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China